CLINICAL TRIAL: NCT04814108
Title: A Phase 2 Open-Label, Multicenter Study to Evaluate Efficacy and Safety of ZN-c3 in Adult Women With Recurrent or Persistent Uterine Serous Carcinoma
Brief Title: A Study of ZN-c3 in Women With Recurrent or Persistent Uterine Serous Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-004
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Uterine Serous Carcinoma
Keywords: uterus; uterine; endometrial; endometrium; serous carcinoma; wee1; Wee-1; usc; Uterine Serous Carcinoma; serous
MeSH Terms: conditions — Cystadenocarcinoma, Serous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZN-c3 Single Agent (Experimental): ZN-c3 (azenosertib) taken orally with food
  Interventions: Drug: ZN-c3

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 is an investigational drug.
  Other Names: azenosertib; KP-2638

SUMMARY:
This is a Phase 2 study to evaluate the clinical activity and safety of ZN-c3 (azenosertib) in adult women with recurrent or persistent uterine serous carcinoma (USC).

DETAILED DESCRIPTION:
This is a Phase 2 open-label, multicenter study to evaluate the clinical activity and safety of ZN-c3 (also known as azenosertib; KP-2638) in adult women with recurrent or persistent uterine serous carcinoma (USC).

ELIGIBILITY:
INCLUSION CRITERIA

1. Females ≥18 years of age at the time of informed consent.
2. Histologically confirmed recurrent or persistent USC for which no other proven effective treatment options are available or any available standard of care therapy was not tolerated or was refused by the subject.

   * Subjects with endometrial carcinoma of mixed histology where the serous component comprises at least 5% of the tumor will be considered eligible.
   * Subjects with carcinosarcomas (even if there is a serous component) are not eligible.
3. Measurable disease per RECIST Guideline Version 1.1
4. Required prior therapy for endometrial cancer:

   1. Treatment with a platinum-based chemotherapy regimen.
   2. Treatment with a PD-(L)1 inhibitor
   3. Known HER2-positive tumors: Treatment with at least 1 HER2-targeted therapy, except for subjects who are not clinically eligible.
5. Adequate hematologic and organ function

EXCLUSION CRITERIA

1. Any of the following treatment interventions within the specified time frame prior to C1D1:

   1. Major surgery within 28 days
   2. Any chemotherapy or targeted tumor therapy within 14 days or 5 half-lives (whichever is shorter).
   3. Radiation therapy within 21 days;
   4. Autologous or allogeneic stem cell transplant within 3 months.
   5. Current use of any other investigational drug therapy <28 days or 5 half-lives (whichever is shorter).
2. Prior therapy with ZN-c3 or any other WEE1 inhibitor, ATR inhibitor, or CHK1/2 inhibitor for USC.
3. A serious illness or medical condition(s) including, but not limited to: Any evidence of bowel obstruction as determined by air/fluid levels on computed tomography (CT) scan, recent hospitalization for bowel obstruction within 3 months prior to C1D1, or recurrent paracentesis or thoracentesis within 6 weeks prior to C1D1.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of TEAEs and incidence of dose modifications | 2 years
  To determine the safety and tolerability of ZN-c3 in subjects with recurrent or persistent USC.
Objective Response Rate as defined by the revised RECIST v1.1 as assessed by ICR | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC

SECONDARY OUTCOMES:
Objective Response Rate as defined by the revised RECIST v1.1. and assessed by ICR and the Investigator. | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC at different doses/schedules
Duration of Response as defined by the revised RECIST v1.1. and assessed by ICR and the Investigator. | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC at different doses/schedules
Progression Free Survival as defined by the revised RECIST v1.1. and assessed by ICR and the Investigator. | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC at different doses/schedules
Clinical Benefit Rate as defined by the revised RECIST v1.1. and assessed by ICR and the Investigator. | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC at different doses/schedules
Time To Response as defined by the revised RECIST v1.1. and assessed by ICR and the Investigator. | 2 years
  To investigate the antitumor activity of ZN-c3 in subjects with recurrent or persistent USC at different doses/schedules

CONTACTS AND LOCATIONS:
Overall Officials: Project Director, Study Director — K-Group Beta (A wholly owned subsidiary of Zentalis Pharmaceuticals)
Locations (52):
- United States (37):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Honor Health, Phoenix, Arizona
  - Arizona Oncology Associates Wilmot HOPE, Tucson, Arizona
  - University of California Irvine Medical Center, Orange, California
  - University of California San Francisco at Mission Bay, San Francisco, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Maryland Oncology Hematology, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - Revive Clinical Research, Sterling, Michigan
  - HCA Midwest Health Kansas City Research, Kansas City, Missouri
  - Center of Hope, Reno, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Optimum Clinical Research Group- Women's Oncology, Albuquerque, New Mexico
  - Westchester Medical Center, Hawthorne, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Trihealth Cancer Institute, Cincinnati, Ohio
  - Ohio State University James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Ascension St. Thomas Midtown Hospital, Nashville, Tennessee
  - Texas Oncology Austin, Austin, Texas
  - Texas Oncology Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology Gulf Coast, Houston, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Health System, Richmond, Virginia
  - Virginia Cancer Specialists, Warrenton, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Icon Cancer Centre- Chermside, Brisbane, Queensland
  - Mater Cancer Care Centre, Mater Misericordiae Limited, Brisbane, Queensland
  - Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Chu de Quebec-Universite, Québec, Quebec
- Georgia (5):
  - LTD High Technology Hospital Medcenter, Batumi, Adjara
  - Rustavi Clinic, Rustavi, Kvemo Kartli
  - Acad. Fridon Todua Medical Center, Tbilisi
  - LTD Innova Medical Center, Tbilisi
  - LTD TIM-Tbilisi Innova of Medicine, Tbilisi